CLINICAL TRIAL: NCT04813406
Title: Anlotinib in Combination With Sintilimab as Second-line Treatment for Advanced Esophageal Squamous Cell Carcinoma (ESCC) : a Multicenter, Single-arm, Open-label Phase Ⅱ Clinical Trial
Brief Title: Study of Anlotinib Plus Sintilimab in the Treatment of Advanced Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-115-02
Record Dates: First submitted 2021-03-21; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — anlotinib; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anlotinib + Sintilimab (Experimental)
  Interventions: Drug: Anlotinib + Sintilimab

INTERVENTIONS:
Drug: Anlotinib + Sintilimab — Anlotinib: 1 capsule (10mg) once a day, d1-d14 per cycle, 3 weeks for a treatment cycle.
  Sintilimab: 200 mg/time, intravenous injection, every 3 weeks is one cycle.

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of anlotinib combined with sindilimab as second-line treatment for advanced esophageal squamous cell carcinoma (ESCC). In addition, we also explored the possible mechanism of anlotinib combined with sindilimab in order to screen out biomarkers that can predict the efficacy of the combination therapy.

DETAILED DESCRIPTION:
China is one of the regions with the highest risk of esophageal cancer in the world, and more than 90% of esophageal cancer is squamous cell carcinoma (SCC). The incidence of esophageal cancer is ranked sixth and the mortality rate ranks fourth in China. At present, the first-line treatment of advanced esophageal cancer is mainly based on the combination of paclitaxel, cisplatin and fluorouracil. After the failure of first-line treatment, there is no standard second-line treatment. The investigators designed a multicenter, single-arm, open-label phase Ⅱ clinical trial of anlotinib combined with sindilimab as second-line treatment for advanced esophageal squamous cell carcinoma (ESCC).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) confirmed diagnosis of esophageal squamous cell carcinoma (excluding mixed type adenosquamous carcinoma )
* Patients undergoing first-line systemic chemotherapy (which may include taxanes, platinum and fluorouracil) progression. For radical concurrent chemoradiotherapy, neoadjuvant/adjuvant therapy (chemotherapy or chemoradiotherapy), if disease progression occurs during treatment or within 6 months after stopping treatment, Count it as a first-line treatment failure.（Note: Patients with advanced or relapsed non target lesions who progress again after radiotherapy alone are included. Palliative treatment for local lesions (non target lesions) lasted for more than 2 weeks.）
* At least one measurable/evaluable lesion by RECIST v1.1（Cavity organ such as esophagus can not be used as measurable lesions）. And the measurable lesions should not have received local treatment such as radiotherapy (The lesion located in the previous radiotherapy area, if confirmed to progress, and meets the RECIST 1.1 standard, can also be used as a target lesion).
* 18~80 years, both men and women.
* Patients who can provide histological specimens for pathological review.
* Eastern Cooperative Oncology Group(ECOG) performance status 0 or 1.
* Life expectancy of ≥ 12 weeks.
* The main organs function normally, that is, the following criteria are met:

  (1) Blood routine examination:
  1. HB≥90g/L;
  2. ANC ≥ 1.5 × 109 / L;
  3. PLT ≥ 80 × 109 / L. (2) Biochemical examination:

     1. TBIL ≤ 1.5ULN
     2. ALT and AST ≤ 2.5ULN
     3. plasma Cr ≤ 1.5ULN or creatinine clearance (CCr) ≥ 60ml / min
     4. left ventricular ejection fraction (LVEF)≥ normal low limit (50%)
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative before enrollment；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped.
* Patients should participate in the study voluntarily and sign informed consent.

Exclusion Criteria:

* The patients who had or were suffering from other malignant tumors within 5 years, except for the cured cervical carcinoma in situ, non melanoma skin cancer and superficial bladder tumor [ta (non-invasive tumor), tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)] and those who developed rapidly within 3 months.
* Patients with a history of perforation and / or fistula within 6 months before the first medication.
* Patients with a high risk of bleeding or perforation due to the apparent invasion of adjacent organs (aorta or trachea) of the esophageal lesion, or patients who have formed fistulas.
* Have received any of the following treatments:

  1. Patients who received Sindilimab therapy or other immunotherapy against PD-1/PD-L1.
  2. Patients who have participated in other drug clinical trials within four weeks.
  3. Enter another clinical study, unless it is an observational (non intervention) clinical study or an intervention clinical study.
  4. Receive the last dose of anticancer treatment (including radiotherapy, etc.) within ≤ 4 weeks before the first use of the study drug.
  5. The patient is using immunosuppressive agents or systemic hormonal therapy for immunosuppression purposes (dose >10 mg/day of prednisone ) and continues to be used within 2 weeks prior to enrollment, except for the use of corticosteroids for local esophageal inflammation and prevention of allergy, nausea and vomiting. In the absence of active autoimmune diseases, inhaled or topical corticosteroids and corticosteroid replacement with a therapeutic dose of prednisone greater than 10 mg / day are permitted.
  6. Patients who had been vaccinated with anti-tumor vaccine or had been vaccinated with live vaccine within 4 weeks before the first administration of the study drug.
  7. The patient had major surgery or severe trauma within 4 weeks before the first use of the study drug.
* A history of immunodeficiency, including a positive HIV test or other acquired, congenital immunodeficiency disease, or a history of organ transplantation.
* The toxicity of previous anti-tumor therapy did not return to ≤ NCI CTC AE v5.01 (except alopecia) or the level specified in the inclusion / exclusion criteria.
* Allergic to monoclonal antibody and anlotinib
* Patients with significant malnutrition. If the patient is receiving intravenous infusion of nutrient solution or requires hospitalization for continuous infusion treatment, then exclusion. Before randomization, patients with good nutrition control for more than 28 days can be enrolled.
* Patients with any severe and / or uncontrolled disease, include:

  1. Patients with hypertension who can not be well controlled by antihypertensive drugs (systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 100 mmHg).
  2. With myocardial ischemia or myocardial infarction, arrhythmia (including QTc ≥ 480ms) and ≥ 2 congestive heart failure (NYHA classification).
  3. Serious or uncontrolled disease or active infection (≥ NCI CTC AE V5.02 infection), which the researchers believe will increase the risk related to research participation, drug delivery or affect the ability of subjects to receive the study drug.
  4. Renal failure requires hemodialysis or peritoneal dialysis.
  5. Poor glycemic control in diabetic patients (FBG > 10mmol / L).
  6. Routine urine showed that urinary protein was ≥ 2+ and 24-hour urinary protein was confirmed to be more than 1.0g.
  7. Patients with epilepsy and need treatment.
* 4 weeks before of enrollment; any sites of bleeding NCI CTC AE grade ≥3, such as unhealed wounds, ulcers or fractures.
* Patients with arteriovenous thrombosis events within 3 months, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism;
* The patient has any active autoimmune disease (such as the following, but not limited to: Interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; patients with vitiligo; complete remission of asthma in childhood, can be included without any intervention after adult, autoimmune hypothyroidism treated with stable dose of thyroid replacement hormone and type I diabetes treated with stable dose of insulin.
* The patient has a history of interstitial lung disease (except radiation pneumonia without hormone therapy) and non infectious pneumonia.
* Patients with active pulmonary tuberculosis infection found by medical history or CT examination, or with a history of active pulmonary tuberculosis infection within one year before enrollment, or with a history of active pulmonary tuberculosis infection more than one year ago but without regular treatment;
* Patients with active hepatitis B (HBV-DNA ≥ 104 copy number / ml or 2000 IU / ml) Or hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the lower limit of detection of the analytical method).
* According to the judgment of the researcher, there are other factors that may cause the subject to be forced to terminate the study, such as suffering from other serious diseases (including mental illness) requiring combined treatment, serious laboratory abnormalities, family or social factors, which may affect the safety of the subject or the collection of experimental data
* Symptomatic central nervous system metastasis and/or cancerous meningitis are known to exist.
* Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | up to 2 year
  From date of randomization until the date of death from any cause

SECONDARY OUTCOMES:
Progress free survival (PFS) | up to 2 year
  From date of randomization until the date of first documented progression or date of death from any cause
Objective Response Rate (ORR) | up to 1 year
  From date of randomization until the date of death from any cause
Disease Control Rate (DCR) | up to 1 year
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD)